CLINICAL TRIAL: NCT05831553
Title: Evaluation of a Tissue Immune Profile (TIP) in Patients Affected by Metastatic TNBC Treated With Upfront Atezolizumab Plus Nab-paclitaxel (TIP)
Brief Title: TIP in Patients Affected by Metastatic TNBC
Acronym: TIP
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Fondazione per la Medicina Personalizzata (Other)
Collaborators: University of Roma La Sapienza (Other)
Responsible Party: Sponsor
Other Study IDs: FMP-2020-01-TIP
Record Dates: First submitted 2023-03-20; First posted 2023-04-26 (Actual); Last update posted 2023-05-06 (Actual); Status verified 2023-05

CONDITIONS: Metastatic Triple-negative Breast Cancer
MeSH Terms: conditions — Triple Negative Breast Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Other
Patient Registry: Yes
Target Follow-Up Duration: 24 Months
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: Tissue Immune Profile — Tissue samples of the patients will be analized for the presence of TILs, CD73 and PDL1 (>=1%)

SUMMARY:
Triple-negative breast cancer (TNBC) is defined by the absence of estrogen receptor (ER), progesterone receptor (PgR), and human epidermal growth factor receptor 2 (HER2) expression on cancer cells. TNBCs accounts for 15-20% of all breast cancers (BC).1 It is characterized by a worse prognosis, increased risk of metastasis to vital organs and a relative lack of therapeutic target if compared to other BC subtypes.2 Therefore, the identification of new molecular targets and therapeutic strategies is a critical need in both early and metastatic setting. TNBC appears to be more immunogenic compared to other BC6. Immunotherapy has recently changed the landscape of therapeutic options in TNBC. Recent clinical trials have shown a significant clinical benefit in patients with metastatic TNBC treated with a combination of chemotherapy and anti PD-1 agents.11-12-13-14-15 In particular, results from IMPASSION 130 trial showed a significant benefit in both progression free survival (PFS) and overall survival (OS) in PD-L1 positive (PD-L1+) patients treated with a combination of atezolizumab and nab-paclitaxel.20 However, about 70% of PD-L1+ patients has experienced a disease progression after one year and about 50% was alive at 2 year. Moreover, no difference in survival endpoint has been seen in PD-L1 negative (PD-L1-) population, with an increase of toxicity and costs related to the addition of a checkpoint-inhibitor. Therefore, the identification of novel biomarkers in addition to PD-L1 and the combination of several biomarkers in a profile with higher predictive capacity is considered an area of urgent clinical need. Some immune-related features that can be identified in tumor microenvironment have been demonstrated to be independent prognostic and predictive factors: TILs, PD-L1, CD73.

1. Tumour-inﬁltrating lymphocytes (TILs) control the clinical progression of various types of cancer7. Breast cancer with higher levels of infiltrating CD8+ cytotoxic T cells have been associated with better patient survival8. Moreover, high levels of stromal CD8+ TILs (sTILs) correlate with higher probability of pCR9. Not only quantitative, but also qualitative analysis of TILs is a promising research area. Some studies suggest that different subtypes of TILs may have an opposite role in tumor microenvironment allowing the induction of both immune activating (es. CD8+) or immune suppressive (es FOXP3+) environment8-9-10.
2. The interaction between programmed cell death protein 1 (PD-1) and its ligand (PD-L1) represents one of the principal mechanisms of immune escape and a therapeutic target for several malignancies13-14. PD-1/PD-L1 interaction attenuates lymphocyte activation and promotes T-regulatory cell development and function, allowing to terminate the immune response15. In breast cancer the prognostic role of PD-1/PD-L1 axis is still uncertain with limited and contrasting data. PD-L1 positivity (≥1%) on immune cells (IC) is the clinical most used threshold, according to the results of IMPASSION 130 trial.18-24
3. Recently, CD73 has been identified as a possible further molecular immunosuppressive target in triple negative breast cancer28. CD73 is expressed on the surface of tumoral cells, stromal cells and immunological cells. By increasing extracellular levels of adenosine monophosphate , CD73 suppresses immune responses. CD73 has been found to be overexpressed in several types of human cancers, and it has been associated with a poor prognosis29-30-31. Particularly Loi et al demonstrated that high CD73 expression is associated with poor prognosis in TNBC and to a low rate of pathological complete response32.

We defined a tissue immune profile positive (TIP+) as the simultaneous presence of TILs≥50%, CD73≤40% and PD-L1≥1%. Any other combination was defined as TIP negative (TIP-) In conclusion, we will evaluate the association between TIP and clinical outcomes (ORR, PFS, OS).

ELIGIBILITY:
Inclusion Criteria:

* Patients able and willing to provide a written informed consent to participate to the study;
* Histological confirmed diagnosis of PD-L1 positive TNBC (> 1%)
* Confirmed radiological or histological diagnosis of metastatic TNBC
* Availability of tumor specimen in order to perform the requested analysis
* Patients eligible for or treated with atezolizumab plus nab-paclitaxel first line as requested for clinical practice
* Availability of complete clinical data on duration, efficacy and safety of the treatment

Exclusion Criteria:

* Sample not sufficient to perform the requested tissue analysis
* Patients unable to provide informed consent or with possible poor compliance with protocol procedures
* Patients with any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule;
* Patients treated with the following drugs, because of the risk of immunosuppression: Chronic or high-dose oral corticosteroid therapy, TNF-inhibitors and Anti-T cell antibodies
* Patients participating in other clinical studies.

Min Age: 18 Years | Sex: Female
Age Groups: Adult, Older Adult
Study Population: Female patients affected by metastatic TNBC (PDL1>1%) treated with upfront atezolizumab plus nab-paclitaxel
Sampling Method: Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-09-16 (Actual); Primary Completion 2025-09-16 (Estimated); Study Completion 2025-09-16 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival | 12 months
  After 12 months from patient enrollment, the presence of disease progression will be assessed

SECONDARY OUTCOMES:
months of Overall Response Rate | through study completion, an average of 1 year
  To evaluate the association between immune profile (TIP) and Objective Response Rate
months of Overall Survival | through study completion, an average of 1 year
  To evaluate the association between immune profile (TIP) and Overall Survival

CONTACTS AND LOCATIONS:
Locations (6):
- Italy (6):
  - Ospedale Santo Stefano, Prato, FI
  - IRCCS Istituto Europeo di Oncologia IEO, Milan, MI
  - Fondazione Policlinico Universitario Agostino Gemelli IRCCS, Roma, RM
  - Azienda Ospedaliero Universitaria Policlinico Umberto I, Roma, RM
  - ospedale Belcolle, Viterbo, VT
  - Istituto Nazionale per lo Studio e la Cura dei Tumori - Fondazione S. Pascale, Napoli